CLINICAL TRIAL: NCT06765018
Title: Tongue Brush (Orabrush) for Reducing Aspiration Pneumonia in Stroke Patients
Acronym: StrOra
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Marburg (Other)
Responsible Party: Principal Investigator, Leona Möller, Leona Möller, MD; Principal Investigator, Consultant in Neurology, University Hospital Marburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-227 BO
Record Dates: First submitted 2024-11-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Dysphagia After Stroke; Aspiration Pneumonias; Ischemic Stroke
Keywords: Dysphagia after stroke; Aspiration Pneumonias; Tongue Coating Index; Bacterial Tongue Colonization; Ischemic Stroke
MeSH Terms: conditions — Pneumonia, Aspiration; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Care Group (No Intervention): Patients in the Routine Care Group receive standard speech therapy during their inpatient stay.
- Tongue Brush Group (Experimental): Patients in the Tongue Brush Group receive standard speech therapy and additionally use the tongue brush twice daily for a period of 3-5 days during their inpatient stay.
  Interventions: Device: Tongue Brush (Orabrush)

INTERVENTIONS:
Device: Tongue Brush (Orabrush) — Patients in this group uses the Tongue Brush (Orabrush) 2 times a day for a duration for 3-5 days until the follow-up-screening takes place.
  Arms: Tongue Brush Group

SUMMARY:
The investigators conduct a controlled prospective experimental intervention study to examine whether the use of a tongue brush (Orabrush) can improve the rate of aspiration pneumonia and dysphagia in patients with ischemic stroke. Secondary outcomes include the impact on bacterial tongue colonization, the Tongue Coating Index, and the length of stay of the patients.The patients will be recruited in the Stroke Unit of the Department of Neurology from November 2024 until approximately October 2026.

DETAILED DESCRIPTION:
As part of a prospective controlled experimental intervention study, patients with ischemic stroke will be recruited in the Stroke Unit of the University Hospital Marburg, who are admitted between November 2024 and approximately October 2026. The primary objective of this study is to investigate the impact of a tongue brush (Orabrush) on the rate of aspiration pneumonia and dysphagia. Secondary outcomes include the analysis of bacterial tongue colonization, the Tongue Coating Index, and the length of stay of the patients. Key study parameters include the aspiration rate, the EAT-10, the GUSS, a tongue swab, and a photograph of the tongue to determine the Tongue Coating Index. Data will be collected on the day of admission and after a duration of 3-5 days. The study has been approved by the relevant ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke and admission on the stroke unit at the University Hospital Marburg
* minimum age: 18 years
* patient is able to consent
* consent has been obtained

Exclusion Criteria:

* surgery in the oral-pharyngeal region
* irradiated patient with a history of tumor in the head and neck region
* missing compliance
* intake of medications with saliva-altering side effects, existing desire to have children, or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Aspiration Pneumonias | From the date of first admission until discharge, with the occurrence of aspiration, within max. 4 weeks pneumonia documented at any point during the inpatient stay.
  Evaluation of the Impact of a Tongue Brush on the Incidence of Aspiration Pneumonia in Patients with Ischemic Stroke.
Severity of dysphagia measured by EAT-10 [score from 0-40] | EAT-10 is assessed on the day of admission and after a period of 3-5 days.
  This study aims to investigate whether the use of a tongue brush has an effect on the severity of dysphagia in ischemic stroke patients compared to the control group. The severity of dysphagia is quantified using the dysphagia screening tool EAT-10. The EAT-10 can have a score ranging from 0 to 40, with the severity of dysphagia increasing as the score rises.
Severity of dysphagia measured by GUSS [score from 0-20] | GUSS is assessed on the day of admission and after a period of 3-5 days.
  This study aims to investigate whether the use of a tongue brush has an effect on the severity of dysphagia in ischemic stroke patients compared to the control group. The severity of dysphagia is quantified using the dysphagia screening tool GUSS. The GUSS can have a score ranging from 0 to 20, with the severity of dysphagia increasing as the score decreases.

SECONDARY OUTCOMES:
Winkel Tongue Coating Index [Score from 0 to 12] | The WTCI of the patients is determined on the day of admission and after 3-5 days.
  Determination of the Winkel Tongue Coating Index (WTCI) in ischemic stroke patients. For this purpose, the tongue is divided into six equal-sized quadrants, and each quadrant is assigned a score from 0 to 2, depending on the severity of tongue coating. In total, a score ranging from a minimum of 0 to a maximum of 12 points can be achieved across the six quadrants. A low score indicates very little tongue coating, while a high score reflects a significant amount of tongue coating.
Microbiological quantification of the tongue's bacterial load through the determination of colony-forming units (CFU) | Bacterial tongue colonization is assessed in the patients through swabbing on the day of admission and after 3-5 days.
  A swab of the tongue is taken from patients with ischemic stroke, and a microbiological quantification of the bacterial load is performed. Depending on the level of CFU, the bacterial load is categorized into the semiquantitative parameters 'low,' 'moderate,' and 'high'.
Length of in-hospital stay in days | Duration of in-hospital stay, measured from the admission date to the discharge date, during the inpatient treatment period. The average length of stay is approximately 6 days, so a maximum time frame of 30 days is chosen for the survey.
  It is investigated how many days patients with ischemic stroke stay in the hospital and whether there is a significant difference in the length of stay between the control and intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No